CLINICAL TRIAL: NCT00412204
Title: A Double-blind, Placebo-controlled, Crossover Study to Evaluate the Effects of Tiotropium Bromide on Gas Exchange in Subjects With COPD During Exercise
Brief Title: Study to Evaluate the Effects of Tiotropium Bromide on Chronic Obstructive Pulmonary Disease (COPD) During Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Gail Gauvreau, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.371
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: COPD
Keywords: double-blind; placebo-controlled; crossover; effects of tiotropium bromide; gas exchange; Chronic Obstructive Pulmonary Disease; exercise.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tiotropium
  Interventions: Drug: tiotropium bromide
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tiotropium bromide — Subjects will be randomized to treatment with tiotropium or placebo. Double-blind medication will be dispensed in HandiHalers to be taken once daily in the morning for 22 days.
  Other Names: tiotropium bromide (Spiriva)
  Arms: 1
Other: Placebo — Subjects will be randomized to treatment with tiotropium or placebo. Double-blind medication will be dispensed in HandiHalers to be taken once daily in the morning for 22 days.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of treatment with tiotropium bromide on efficiency of gas exchange and exercise performance in COPD subjects during exercise.

DETAILED DESCRIPTION:
This study will investigate the effect of tiotropium on gas exchange during exercise. In addition, we hypothesize that bronchodilation by tiotropium will open functional lung units improving gas exchange in subjects with COPD. While other studies have shown that tiotropium improves exertional dyspnea and exercise tolerance, and reduces resistive and elastic work in subjects with COPD, there have been no investigations of the effects of anti-cholinergic bronchodilation on gas exchange. This study will confirm and extend earlier observations on exertional dyspnea and exercise tolerance.

Efficiency of gas exchange will be evaluated through assessments of metabolic demand (VO2) cardiac output (Q), ventilation (V) in overall terms i.e. Q/VO2, V/VO2.

Improved efficiency of gas exchange will reduce the ventilatory demand for a given workload, providing an alternate mechanism for the observed improvement in exertional dyspnea and exercise tolerance in subjects with COPD. The overall ventilation required to meet metabolic demands is dependent on the alveolar volume which can be easily measured using inert gases. This is conveniently measured during the DLco maneuver which will be measured. In general, ventilation increases with metabolic demand but increases progressively as the VA and KCO decline in patients with COPD. These factors may be amenable to improvement using anticholinergic agents. In addition the recruitment of additional alveolar volume provides an additional pathway for blood flow through the lung increasing overall cardiac output and enhancing the responsiveness of peripheral muscle in these patients. These have not been considered and exploited as potential therapeutic goals.

Study Evaluations:

Treatment Period: Visits 2, 3, 5 and 6

* Vital signs (seated)
* 12 lead ECG
* Medication washout compliance.
* Stage one exercise test (refer to section 11.1.7)
* Randomization will occur at Visit 2.
* At visit two the subject will be trained in the use of a HandiHaler
* Study medication will be dispensed at Visit 2 and 5
* Administer study medication (Visits 2,3,4,5 and 6)

Treatment Period: Visits 4 and 7

* Vital signs (seated)
* Administer study medication
* Constant load exercise test (refer to section 11.1.8)
* Collect study medication
* Medication accountability
* Adverse event (A follow up visit must be scheduled if there are any ongoing AEs at visit 7)

Follow up Visit (within 30 days of visit 7):

This visit will take place only if clinically significant abnormalities are seen after all results from Visit 7 are obtained and reviewed by the Investigator and Medical Monitor.

After informed consent, patients will attend an initial screening visit (Visit 1) for review of medical history, clinical assessment, complete pulmonary function testing (plethysmography and spirometry). A symptom-limited incremental cycle exercise test, with measurement of incremental and peak VO2, carbon dioxide output (VCO2), minute ventilation (Ve), Vt, respiratory frequency, heart rate (HR), oxyhemoglobin saturation by pulse oximeter (SpO2) and modified Borg score for breathlessness will also be performed at screening, as well as measurements of airway responses to salbutamol.

Patients who meet the eligibility requirements will be randomized to treatment with tiotropium or placebo. Double-blind medication will be dispensed in HandiHalers to be taken once daily in the morning for 22 days. Patients will report to the laboratory for two separate treatment periods with a washout of 4-6 weeks between treatment periods. A patient diary card will be kept to document morning doses of study medication for calculation of compliance. The patient will return used medication capsules for confirmation of medication compliance. Safety will be assessed by examining adverse events (AEs), resting and exercise electro cardio grams (ECG's), routine laboratory tests and vital signs.

In the event of treatment of an exacerbation with oral corticosteroids, any scheduled visit will be delayed for 1 week following the last dose of steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be current or ex-smokers with a cigarette smoking history of > 10 pack years.
* All patients must have a diagnosis of COPD.
* Patients maintained on a daily dose of inhaled corticosteroids need to be at a constant dose at 4 weeks prior to study entry.

Exclusion Criteria:

* Patients with significant diseases other than COPD.
* Patients with a history of a recent (i.e. six months or less) myocardial infarction.
* Patients with unstable or life threatening cardiac arrhythmias including any patient with a newly diagnosed, clinically relevant arrhythmia on the ECG performed on Visit 1.
* Patients who have been hospitalized for heart failure (NYHA class III or IV) within the past year.
* Patients with a history of life threatening pulmonary obstruction, or history of cystic fibrosis or clinically evident bronchiectasis.
* Patients who have undergone thoracotomy with pulmonary resection.
* Patients with any respiratory infection or exacerbation in the six weeks prior to Visit 1.
* Patients who regularly use daytime oxygen therapy for more than one hour per day and who in the investigator's opinion, will be unable to abstain from the use of oxygen therapy during testing.
* Patients who are currently in a pulmonary rehabilitation program or who have completed a pulmonary rehabilitation program within four weeks of Visit 1.
* Patients with known active tuberculosis.
* Patients with a history of cancer within the past five years.
* Pregnant or breastfeeding women or women of childbearing potential not using a medically approved means of contraception.
* Patients with known hypersensitivity to anti-cholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
* Patients with a history of significant alcohol or drug abuse in the previous year.
* Patients with have taken an investigational drug within 30 days or 6 half lives (whichever is greater) prior to Visit 1.
* Patients using oral corticosteroid medication and unstable doses (i.e. less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg prednisone per day or 20 mg every other day.
* Patients who use rescue medication (Salbutamol) more than 8 puffs/day.
* Patients who have used tiotropium (Spiriva) within 4 weeks prior to Visit 1.
* Patients who have frequent exacerbations which could be expected to interfere with participation in the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficiency of gas exchange Ve/VO2 and Ve/VCO2 before and after 3 weeks treatment with tiotropium compared to placebo. | Before and after 3 weeks treatment with tiotropium compared to placebo.

SECONDARY OUTCOMES:
Intensity of dyspnea | Before and after 3 weeks treatment with tiotropium compared to placebo.
Effort during incremental and steady state exercise | Before and after 3 weeks treatment with tiotropium compared to placebo.
Exercise endurance capacity | Before and after 3 weeks treatment with tiotropium compared to placebo.
Dyspnea and leg effort | Before and after 3 weeks treatment with tiotropium compared to placebo.
Ventilatory capacity | Before and after 3 weeks treatment with tiotropium compared to placebo.
Alveolar volume | Before and after 3 weeks treatment with tiotropium compared to placebo.
Kco | Before and after 3 weeks treatment with tiotropium compared to placebo.
Cardiac output at rest and during steady state exercise before and after 3 weeks treatment with tiotropium compared to placebo. | Before and after 3 weeks treatment with tiotropium compared to placebo.
Ventilation/perfusion before and after 3 weeks treatment with tiotropium compared to placebo | Before and after 3 weeks treatment with tiotropium compared to placebo.
Ventilation during incremental and steady state exercise before and after 3 weeks treatment with tiotropium compared to placebo. | Before and after 3 weeks treatment with tiotropium compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University; Keiran Killian, MD, Study Director — McMaster University